CLINICAL TRIAL: NCT04012879
Title: Study Evaluating the Efficacy and Safety With CD19CAR-T for Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, Li Yu, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ALL001-CART
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Relapsed Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): After 6 days of pre-chemotherapy, patients in study group will be injected with CD19CART cell at the dose of 5×10^4 cells/kg in 36-96 hours
  Interventions: Combination Product: CD19 CART

INTERVENTIONS:
Combination Product: CD19 CART — CD19 CART

SUMMARY:
This study is a single-arm, open label, phase I clinical trial to evaluate the safety and feasibility of CD19CAR-T in treatment of relapsed / refractory acute lymphoblasic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with Relapsed or refractory acute lymphocyte leukemia with CD19 positive
2. Age 18 to 65 years old, both male and female;
3. Is expected to survive more than 12 weeks;
4. Physical condition is good: 0-1 score ECOG score;
5. No obvious abnormal heart, liver, kidney, no large wounds that haven't healed on the body;
6. Into groups to participate in voluntarily, good adherence, can cooperate test observation, childbearing age women must be 7 days before starting treatment expert pregnancy test and the results were negative, and signed a written informed consent form.

Exclusion Criteria:

1. Organ failure, such as heart: Class III and IV; liver: to Child grading of liver function grade C; kidney: kidney failure and uremia stage; lung: symptoms of severe respiratory failure; brain: disorder of consciousness;
2. Existing serious acute infection, uncontrollable, or have fester sex and chronic infection, wound in delay no more;
3. Pregnancy and lactation women;
4. Patients who have participated in other clinical trials or other clinical trials in the past 30 days;
5. The Investigator believe the patients should not participate in this experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
recovery rate of patients being treated with CD19CAR-T | 6 months
  the recovery rate of patients consists of complete recovery rate and partial recovery rate of patients being treated with CD19 CAR-T

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen University General Hospital, Shenzhen, China